CLINICAL TRIAL: NCT04347616
Title: Infusion of ex Vivo-generated Allogeneic Natural Killer Cells in Combination With Subcutaneous IL-2 in Patients With Acute Myeloid Leukemia: a Phase I/IIa Study
Brief Title: Natural Killer-cell Therapy for Acute Myeloid Leukemia
Acronym: NK4AML
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEMAML42; 2019-001929-27 (EudraCT Number)
Record Dates: First submitted 2020-04-06; First posted 2020-04-15 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia, Relapsed, Adult
Keywords: Natural Killer cells; Acute Myeloid Leukemia; Cellular Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Intervention Model Description: The study is divided in two phases. In phase I, we will determine the safety of our UCB-NK cell product with or without sc IL-2, following a non-myeloablative immunosuppressive conditioning regimen in patients with AML. Three patients will receive NK cells without IL-2. If no dose limiting toxicities occur another three patients will receiving NK cells with a low dose IL-2, and if safe, another six patients will receive NK cells with a higher dose IL-2.
  The primary objective of phase IIa of the study is to evaluate the effect of UCB-NK cell adoptive immunotherapy in combination with SC IL-2 following a non-myeloablative immunosuppressive conditioning regime on disease activity in patients with AML. Therefore 17 patients will be evaluated using a Simon's optimal two-stage single-arm study design, with 10 patients in the first stage and an additional 7 patients in the second stage. These patients will receive NK cells with the highest tolerable dose IL-2, established after phase I.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NK cells without IL-2 (Experimental): On day 0, patients will receive a fixed dose of 1.0-3.0 x 10^9 allogeneic UCB-NK cells. Prior to NK cell infusion, patients will receive cyclophosphamide and fludarabine (Cy/Flu) based lymphodepleting chemotherapy. NK cells administration will not be followed by sc IL-2. N=3.
  Interventions: Biological: UCB-NK cells
- NK cells with low dose IL-2 (Active Comparator): On day 0, patients will receive a fixed dose of 1.0-3.0 x 10^9 allogeneic UCB-NK cells. Prior to NK cell infusion, patients will receive cyclophosphamide and fludarabine (Cy/Flu) based lymphodepleting chemotherapy. IL-2 will be administered in a fixed dose of 3.0 x 10^6 units starting 4 hours after NK cell infusion and given every other day for 6 doses in total. N=3
  Interventions: Biological: UCB-NK cells; Drug: IL-2
- NK cells with higher dose IL-2 (Active Comparator): On day 0, patients will receive a fixed dose of 1.0-3.0 x 10^9 allogeneic UCB-NK cells. Prior to NK cell infusion, patients will receive cyclophosphamide and fludarabine (Cy/Flu) based lymphodepleting chemotherapy. IL-2 will be administered in a fixed dose of 6.0 x 10^6 units starting 4 hours after NK cell infusion and given every other day for 6 doses in total. N=6
  Interventions: Biological: UCB-NK cells; Drug: IL-2

INTERVENTIONS:
Biological: UCB-NK cells — Natural killer cells generated from CD34+ hematopoietic progenitor cells derived from an allogeneic umbilical cord blood
Drug: IL-2 — In vivo cytokine support
  Other Names: Aldesleukin
  Arms: NK cells with higher dose IL-2; NK cells with low dose IL-2

SUMMARY:
This study investigates an innovative treatment for relapsed or refractory acute myeloid leukemia exploiting administration of ex vivo-generated allogeneic natural killer (NK) cells with preceding non-myeloablative conditioning chemotherapy with or without subsequent in vivo IL-2 cytokine support.

DETAILED DESCRIPTION:
This study investigates an innovative treatment for relapsed or refractory acute myeloid leukemia (AML) exploiting administration of ex vivo-generated allogeneic natural killer (NK) cells with preceding non-myeloablative conditioning chemotherapy with or without subsequent in vivo IL-2 cytokine support.

This is a prospective phase I/IIa study. The first phase is a IL-2 dose-escalating safety study in twelve patients. The second phase of the study is designed as a Simon's optimal two-stage single-arm phase IIa study, comprising seventeen patients. Prior to NK cell infusion, all patients will receive cyclophosphamide and fludarabine (Cy/Flu) based lymphodepleting chemotherapy. On day 0, all patients will receive a fixed dose of 1.0-3.0 x 10^9 allogeneic umbilical cord blood-derived NK cells (UCB-NK cells). These cells are generated ex vivo from CD34+ hematopoietic progenitor cells obtained from an allogeneic UCB unit.

In phase I of the study patients will receive UCB-NK cells without subcutaneous (SC) IL-2, with lower dose SC IL-2 or with higher dose SC IL-2 (n=3 per treatment group, n=6 in the highest tolerable dose). After establishing the safety of UCB-NK cells combined with SC IL-2, we will continue with phase IIa of the study, with ten patients in the first stage (including the six patients from phase I with comparable IL-2 dose) and if clinical efficacy is achieved an additional seven patients in the second stage.

ELIGIBILITY:
Inclusion Criteria:

* AML patients (de novo and secondary) or patients with MDS excess blasts-2 according to WHO criteria 2016, who have stable disease or non-rapidly progressive disease with or without disease controlling medication who are (at time of inclusion) ineligible for allo-SCT.
* Patients may belong to any of the following categories:

  * Relapsed/refractory disease after treatment with intensive chemotherapy, hypomethylating agents, targeted agents, autologous or allo-SCT (at least 6 months ago) and DLI
  * Newly diagnosed, untreated patients ineligible for allo-SCT

Other inclusion criteria:

* Age ≥ 18 years
* WHO performance 0-2
* Life expectancy of > 4 months
* Written informed consent
* Hydrea is allowed as pre-treatment to control blast count until day -3
* Other disease controlling medication is allowed until day -7

Exclusion Criteria:

* Progressive disease according to ELN criteria in case of previous therapy
* Patients on immunosuppressive drugs or active GvHD
* Patients with active infections (viral, bacterial or fungal); acute anti-infectious therapy must have been completed within 14 days prior to study treatment
* Severe cardiovascular disease (CTCAE III-IV)
* Severe pulmonary dysfunction (CTCAE III-IV)
* Severe renal dysfunction (CTCAE III-IV)
* Severe hepatic dysfunction (CTCAE III-IV)
* Severe neurological or psychiatric dysfunction (CTCAE III-IV)
* Patients on concurrent chemotherapy or interferon-alpha treatment
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Evaluate Safety and Toxicity using the CTCAE toxicity criteria | 28 days
  Patients will be evaluated intensively using the CTCAE toxicity criteria and graft versus host disease (GvHD) classification criteria, defining dose limiting toxicities (DLTs): 1. Any treatment-emergent non-hematologic grade 3 toxicity lasting >72 hours, except for transient constitutional symptoms, diarrhea, fatigue or skin rash not requiring systemic steroid therapy. 2. Acute GvHD >grade 2 within 6 weeks of the first IL-2 dose. If in any of the three patients of each individual cohort of the phase I study a DLT occurs, the cohort will be extended to 6 patients. If 2 patients experience DLT within a cohort of 3 or 6 patients the study will be stopped in case the patients were only receiving NK cells or the study will be continued without IL-2 or the lower dose of IL-2 in case the patients were receiving NK cells in combination with IL-2. Serious, life threatening adverse events or grade 4 toxicity will be a reason to terminate the study or continue without IL-2 cytokine support.
Phase IIa: % blasts or % minimal residual disease (MRD) in the bone marrow | 28 days
  The primary objective of phase IIa of the study is to evaluate the effect of UCB-NK cell adoptive immunotherapy in combination with SC IL-2 following a non-myeloablative immunosuppressive conditioning regime on disease activity in patients with AML. At day 28 a bone marrow biopsy will be performed to evaluate % blasts or % minimal residual disease (MRD) in the bone marrow. A complete remission is defined as BM blasts <5%; marrow should not be merely 'aplastic': at least 200 cells should be enumerated or cellularity should be at least 10%. MRD will be evaluated by flow cytometry (leukemia associated phenotypes (LAPs)) and/or molecular quantification of patient specific mutations (PCR).
  For phase IIa of the study the clinical evaluation data (% blasts and % MRD positivity) will be translated in a clinical response (stable disease, partial remission, complete remission) and quantitative presented.

SECONDARY OUTCOMES:
Evaluation of the in vivo lifespan and expansion potential of the NK cells following adoptive transfer and IL-2 administration. | 28 days
  We will determine the percentage and absolute number of donor-derived NK cells in peripheral blood and bone marrow after infusion using flow cytometry and DNA chimerism analysis. A positive expansion rate of the infused NK cells requires an absolute number of ≥100 donor-derived NK cells per μl blood at day +7 and/or +14.
Exploration of the functional activity of the donor NK cells in PB and BM, with or without SC IL-2 administration. | 28 days
  NK cells from peripheral blood and bone marrow will be obtained. These cells will be stimulated in vitro for 4 hours and subsequently the degranulation marker CD107a and immunoregulatory marker IFNy will be measured by flow cytometry. These results can be compared between patients that did receive IL-2 or did not.
Evaluation of plasma cytokine concentrations (IL-2, IL-15, IL-7, IFN-γ, TNFα, IL-6) pre- and post-infusion of IL-2. | 28 days
  This will be correlated with absolute lymphocyte count and in vivo NK cell persistence and expansion.
Number of patients eligible for allo-SCT based on hematologic response | 28 days
  Only in Phase IIa.

CONTACTS AND LOCATIONS:
Overall Officials: N.P.M. Schaap, Principal Investigator — Department of Hematology
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dolstra H, Roeven MWH, Spanholtz J, Hangalapura BN, Tordoir M, Maas F, Leenders M, Bohme F, Kok N, Trilsbeek C, Paardekooper J, van der Waart AB, Westerweel PE, Snijders TJF, Cornelissen J, Bos G, Pruijt HFM, de Graaf AO, van der Reijden BA, Jansen JH, van der Meer A, Huls G, Cany J, Preijers F, Blijlevens NMA, Schaap NM. Successful Transfer of Umbilical Cord Blood CD34+ Hematopoietic Stem and Progenitor-derived NK Cells in Older Acute Myeloid Leukemia Patients. Clin Cancer Res. 2017 Aug 1;23(15):4107-4118. doi: 10.1158/1078-0432.CCR-16-2981. Epub 2017 Mar 9. PMID 28280089